CLINICAL TRIAL: NCT02067884
Title: Real Time Contrast Enhanced Ultrasound and Ultrasound-Based Elastography: Novel Techniques in Assessment of Treatment Response to Neoadjuvant Chemotherapy for Breast Cancer
Brief Title: Contrast Enhanced Ultrasound and Shear Wave Elastography in Measuring Response in Patients With Breast Cancer Receiving Chemotherapy Before Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); L K Whittier Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1B-13-8; NCI-2014-00085 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-13-8 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2014-02-04; First posted 2014-02-20 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (CEUS, SWE) (Experimental): Patients undergo dynamic contrast-enhanced ultrasound imaging and shear wave elastography at baseline, 2-3 weeks after initiation of chemotherapy, and before surgery.
  Interventions: Procedure: dynamic contrast-enhanced ultrasound imaging; Procedure: shear wave elastography; Drug: Definity, (Lipid Microspheres) Intravenous Suspension; Device: Philips Shear Wave Elastography

INTERVENTIONS:
Procedure: dynamic contrast-enhanced ultrasound imaging — Undergo CEUS
  Other Names: DCE-USI
Procedure: shear wave elastography — Undergo SWE
  Other Names: SWE
Drug: Definity, (Lipid Microspheres) Intravenous Suspension — Participant will receive contrast agent by intravenous administration
  Other Names: Perflutren Lipid Microsphere
Device: Philips Shear Wave Elastography — Equipment used for SWE
  Other Names: Shear Wave Elastography

SUMMARY:
This pilot clinical trial studies contrast enhanced ultrasound and shear wave elastography in measuring response in patients with breast cancer receiving chemotherapy before surgery. New imaging procedures, such as contrast enhanced ultrasound and shear wave elastography, may predict treatment response earlier and more accurately than contrast enhanced magnetic resonance imaging.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish a quantitative prediction rule for accurate and early prediction of the pathologic tumor response assessed post-surgery, using the change of contrast enhanced ultrasound (CEUS) assessed tumor size and perfusion characteristics before (baseline) and 2-3 weeks following initiation of neoadjuvant chemotherapy (NAC).

II. To assess the agreement between CEUS based classification rule and pathologically determined treatment response (baseline versus pre-surgical scan).

III. To establish a quantitative prediction rule for accurate and early prediction of the pathologic tumor response assessed post-surgery, using the change in propagation velocity of a shear mechanical wave in tissue before (baseline) and 2-3 weeks following initiation of NAC.

IV. To assess the agreement between shear wave elastography (SWE) based classification rule and pathologically determined treatment response (baseline versus pre-surgical scan).

SECONDARY OBJECTIVES:

I. To explore the role of combined CEUS + SWE features obtained at early treatment phase (2-3 weeks following initiation of NAC), in accurately predicting the pathologically determined tumor response.

II. To investigate the agreement in assessment of therapy response to NAC between CEUS versus contrast enhanced magnetic resonance imaging (CE MRI) and SWE versus CE MRI for baseline versus pre-surgery scan and to identify discordant cases using scatter plot and contingency tables.

OUTLINE:

Patients undergo dynamic contrast-enhanced ultrasound imaging and shear wave elastography at baseline, 2-3 weeks after initiation of chemotherapy, and before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed breast cancer (by core needle biopsy)
* Women with >= 2 cm clinically or radiologically measureable breast cancer
* Women scheduled to receive neoadjuvant chemotherapy as part of their treatment plan
* Women competent to sign study specific written Informed Consent
* Women willing to comply with protocol requirements

Exclusion Criteria:

* Women who are pregnant
* Women who have undergone open surgical (excisional) biopsy for breast cancer diagnosis
* Women who have had a prior history of breast cancer in the same breast
* Women with known cardiac shunt, pulmonary hypertension or hypersensitivity to perflutren agent
* Women who cannot consent for themselves

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-12-19 (Actual); Primary Completion 2016-09-25 (Actual); Study Completion 2016-09-25 (Actual)

PRIMARY OUTCOMES:
Model predicted treatment response for CEUS and SWE | Up to 1 year
  Weighted Kappa will be used to assess the agreement.
Pathologically determined treatment response for CEUS and SWE | Up to 1 year
  Weighted Kappa will be used to assess the agreement.

SECONDARY OUTCOMES:
Treatment response predicted by novel ultrasound techniques | Up to 1 year
  Weighted Kappa will be used to assess the agreement. Scatter plots and contingency tables will be used to identify discordant cases between US techniques and CE MRI.
Treatment response predicted by CE MRI | Up to 1 year
  Weighted Kappa will be used to assess the agreement. Scatter plots and contingency tables will be used to identify discordant cases between US techniques and CE MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Hovanessian-Larsen, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States